CLINICAL TRIAL: NCT05375578
Title: Urdu Translation and Cross Cultural Validation of Wayfinding Questionnaire for Stroke Patients
Brief Title: Urdu Translation of Wayfinding Questionnaire for Stroke Patients
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/Lhr/22/0207 Suhair Asif
Record Dates: First submitted 2022-04-28; First posted 2022-05-16 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Stroke
Keywords: Way finding Questionnaire, Navigation, Cognition.
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Descriptive analytical study to translate WQ in Urdu Language. The WQ is in English Language the name of the author of WQ is Van der Ham Et al and firstly introduced in 2013. The reliability of this English tool is 0.70 to 0.80 it has been translated in various Languages i.e Hungarian, Dutch and Chinese and suffering from stroke. But it was not translated in Urdu Language. No such study has been previously conducted in Pakistan region which translates the scale and follows the proper cross-cultural adaptation

DETAILED DESCRIPTION:
For resolving such problem WQ play pivotal role in accessing navigation problem of stroke patients it is a very reliable tool for accessing navigation issue. The scale consists of 22 items. All the items dated from 01 to 07 in which stroke patients are accessed. The patients who are taken in the study age from 18 to 65 years. As the WQ is a well-developed measurement scale for accessing navigation in stroke patients. It is meaningful to validate its Urdu version. The translation and cultural adaptation process would start after obtaining approval from the developer of the original WQ. This would be done according to bitten guidelines. The purpose will be to gain uniformity in the translation of both the target Language and source Language. This will involve 5 steps which is forward translation, synthesis 1, back translation, synthesis 2 and pallet testing. The second step would be done according to the Beaton guidelines in which psychometric properties will be measured that is internal consistency, test retest reliability, Discriminant validity, Convergent Validity, Content Validity and Factor analysis

ELIGIBILITY:
Inclusion Criteria:

* Age group 45-65 years
* Male and Female.
* Both ischemic and hemorrhagic stroke
* Patient may have First or Recurrent Stroke.
* Recovery is > 6 months of First Stroke event
* MMSE score > 25

Exclusion Criteria:

* Population suffering from Severe Global Aphasia.
* Population suffering from Severe Mobility Problem.
* Any other neurological disease dementia
* Alzheimer's
* Cognitive Decline before Stroke

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stroke
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Wayfinding Questionnaire | 8 months
  For resolving such problem WQ play pivotal role in accessing navigation problem of stroke patients it is a very reliable tool for accessing navigation issue. The scale consists of 22 items. All the items rated from 1 to 7 in which stroke patients are assessed. The patients who are taken in the study age from 45 to 65 years.

SECONDARY OUTCOMES:
Reliability of translated version of WQ | 8 months
  To determine the reliability of cross-culturally adapted and translated WQ in the patients with stroke.
  Reliability or reproducibility reference to a measure to produce the same results when administered at to intervals between different visits of the patients. Thus this will be measured through test re-test reliability
Validity of translated version of WQ | 8 months
  To determine the validity of cross-culturally adapted and translated WQ for stroke patients in Urdu language

CONTACTS AND LOCATIONS:
Overall Officials: Tehreem Mukhtar, Principal Investigator — Riphah International University
Locations (1):
- Hospital, Lahore, Pakistan(Punjab_, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamre C, Fure B, Helbostad JL, Wyller TB, Ihle-Hansen H, Vlachos G, Ursin MH, Tangen GG. Impairments in spatial navigation during walking in patients 70 years or younger with mild stroke. Top Stroke Rehabil. 2020 Dec;27(8):601-609. doi: 10.1080/10749357.2020.1755814. Epub 2020 Apr 21. PMID 32316862
- [Background] de Rooij NK, Claessen MHG, van der Ham IJM, Post MWM, Visser-Meily JMA. The Wayfinding Questionnaire: A clinically useful self-report instrument to identify navigation complaints in stroke patients. Neuropsychol Rehabil. 2019 Aug;29(7):1042-1061. doi: 10.1080/09602011.2017.1347098. Epub 2017 Jul 18. PMID 28720024